CLINICAL TRIAL: NCT02077114
Title: Peptide Vaccination in Combination With Either Ipilimumab or Vemurafenib for the Treatment of Patients With Unresectable Stage III or IV Malignant Melanoma A Phase I Study (First in Man)
Brief Title: Vaccination With Peptides in Combination With Either Ipilimumab or Vemurafenib for the Treatment of Unresectable Stage III or IV Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Jon Bjørn, MD, Herlev Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM1304
Record Dates: First submitted 2014-02-20; First posted 2014-03-04 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Malignant Melanoma With Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ipilimumab (Experimental): Patient who according to standard criteria are candidates to treatment with Ipilimumab
  Interventions: Biological: Vaccine consisting of a peptide derived from the protein IDO
- Vemurafenib (Experimental): Patients who according to standard criteria are candidates to treatment with Vemurafenib
  Interventions: Biological: Vaccine consisting of a peptide derived from the protein IDO

INTERVENTIONS:
Biological: Vaccine consisting of a peptide derived from the protein IDO — All patients will receive seven vaccines containing IDOlong
  Other Names: IDOlong

SUMMARY:
The purpose of the study is to assess whether a vaccine containing a small fragment of the protein IDO, which may be present in cancer cells and cells of the immune system, is safe to use in combination with either Ipilimumab or Vemurafenib in the treatment of malignant melanoma that has metastasized.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria - all patients

  1. Age ≥ 18
  2. Measurable disease according to RECIST 1.1
  3. ECOG performance status ≤ 2
  4. Patients with asymptomatic brain metastases allowed (treatment with systemic glucocorticoids is not compatible with participation)
  5. Women of childbearing potential must have negative s-hCG prior to initiation of treatment, and use effective contraception during treatment and up to 26 weeks after the last treatment. Safe contraception include: Birth control pills, intrauterine devices, depot injection of progesterone, subdermal implantation (eg Implanon), hormonal vaginal ring and transdermal patch.

All patients must meet all inclusion criteria in the treatment group they belong to.

Inclusion criteria Vemurafenib and peptide vaccine

1. Histologic confirmed stage III (non-operable) or stage IV melanoma with BRAF V600 documented mutation
2. Patients should be fully recovered from any previous systemic or topical treatment for metastatic malignant melanoma
3. Adequate haematological, renal and hepatic function:

   * Neutrophils ≥ 1.5 x 10^9 / l
   * Platelet count ≥ 100 x 10^9 / l
   * Hemoglobin ≥ 5.6 mmol / l
   * Serum creatinine ≤ 1.5 times upper normal limit
   * AST or ALT ≤ 2.5 times upper normal limit (≤ 5 times upper normal limit if it is considered that an increase due to liver metastases)
   * Serum bilirubin ≤ 1.5 times upper normal limit
   * Alkaline phosphatase ≤ 2.5 times upper normal limit (≤ 5 times upper normal limit if it is considered that an increase due to liver metastases)

Inclusion criteria Ipilimumab and peptide vaccine

1. Histologic verified stage III (non-operable) or stage IV malignant melanoma
2. Patients previously treated with anti-CTLA-4 therapy can be included, unless this treatment is stopped due to lack of efficacy or side effects
3. There must be at least 21 days since last systemic treatment of malignant melanoma and the patient must be free of side effects from this treatment. After palliative radiotherapy elsewhere than in the brain, treatment with Ipilimumab and peptide vaccine can be initiated, without a 21 day break. When radiotherapy is used for brain metastases, treatment, however, can only be initiated when the patient is not dependent on prednisolone.
4. Adequate haematological, renal and hepatic function:

   * Leukocytes ≥ 2 x 10^9 / l
   * Neutrophils ≥ 1 x 10^9 / l
   * Platelet count ≥ 75 x 10^9 / l
   * Hemoglobin ≥ 5.6 mmol / l (possibly after transfusion)
   * Serum creatinine ≤ 2 times upper limit of normal
   * AST or ALT ≤ 2.5 times upper normal limit (≤ 5 times upper normal limit if it is considered that an increase due to liver metastases)
   * Serum bilirubin ≤ 2 times upper normal limit (except for patients with Gilbert's syndrome, which allowed bilirubin up to 3.0 mg / dL)

Exclusion Criteria:

* Exclusion criteria - all patients

  1. Concomitant immunosuppressive therapy including prednisolone and methotrexate
  2. Known infection with HIV, hepatitis B and C virus, even if infection remain stable with medical treatment
  3. Other malignancy within the past three years, other than squamous cell and basal cell skin carcinoma
  4. Serious somatic disease, severe asthma, severe COPD, poorly controlled cardiovascular disease or diabetes
  5. Patients must not have undergone major intestinal surgery within the last 28 days.
  6. Severe allergies or previous anaphylactoid reactions
  7. Pregnant or lactating women
  8. Psychiatric illness that is perceived by the investigator to likely affect patient compliance
  9. Known hypersensitivity to ingredients in the adjuvant substances Montanide or Aldara cream

Exclusion Criteria Vemurafenib and peptide vaccine

1. At least one of the following within the past six months: myocardial infarction, severe / unstable angina pectoris, symptomatic congestive heart failure, cerebrovascular event or transient ischaemic attack, pulmonary embolism, poorly controlled hypertension,
2. Congenital long QT syndrome, previous or current significant ventricular or atrial dysrhythmia ≥ 2nd degree (NCI CTCAE version 4.0)
3. Corrected QT interval ≥ 450 msec at baseline
4. Uncontrolled medical illness such as infection requiring intravenous antibiotics
5. Other severe acute, chronic or psychiatric condition or abnormal laboratory value, which can increase the risk associated with Vemurafenib treatment

Exclusion Criteria Ipilimumab and peptide vaccine

1. Autoimmune diseases: History of inflammatory bowel disease, including Crohn's disease and ulcerative colitis, systemic autoimmune disease eg. rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis, including Wegener granulomatosis. Patients with motor neuropathy believed to be of autoimmune origin such as Guillain-Barre and Myasthenia gravis can not be included in the study.
2. Treatment with any vaccine to prevent infection within 28 prior to initiation of treatment with the peptide vaccine and Ipilimumab
3. Systemic treatment with prednisolone.
4. Life-threatening diseases that require treatment with immunosuppressive agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events during and after treatment as a Measure of Safety and Tolerability. | Ipilimumab+vaccine combination: Day 84. Vemurafenib+vaccine combination: Day 56.
  Primary endpoints will be assessed according to CTCAE ver. 4.0

SECONDARY OUTCOMES:
Vaccine related immune response | Ipilimumab: Day 1 (before first treatnent), day 21, day 42, day 63 and at day 84. Thereafter every 12 weeks until progression or up to 104 weeks. Vemurafenib: Day 1, day 28, day 56. Thereafter every 28 days until progression or up to week 104 weeks.
  Reactivity towards epitopes nested within the sequence of the peptide used for vaccination, will be assessed in T cells from peripheral blood, obtained at the specified sample times. Reactivity will be assessed using ELISpot technology, where secretion of interferon gamma and tumor necrosis factor alpha is measured during in vitro stimulation with the peptide used for vaccination. In addition to this, combinatorial coding with fluor chrome conjugated HLA tetramers are used to enumerate precursor frequency of CD8 T cells specific for epitopes within the peptide sequence

CONTACTS AND LOCATIONS:
Overall Officials: Jon Bjørn, MD, Principal Investigator — Center for Cancer Immune Therapy; Inge Marie Svane, MD, PhD, Professor, Study Chair — Center for Cancer Immune Therapy
Locations (1):
- Department of Oncology, Herlev Hospital, Herlev, Denmark

REFERENCES:
- See also: Related Info — http://www.herlevhospital.dk/ccit-denmark/menu/